CLINICAL TRIAL: NCT01047020
Title: Motor Proficiency And Physical Activity in Adult Survivors of Childhood ALL
Brief Title: Motor Proficiency And Physical Activity in Adult Survivors of Childhood Acute Lymphoblastic Leukemia (ALL)
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Tennessee (Other); University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: MTRPAL; R01CA132901 (NIH)
Record Dates: First submitted 2010-01-08; First posted 2010-01-12 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Impairments of musculoskeletal Health;; Physical activity;; Motor Proficiency;
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ALL survivors: The study sample for this research will be recruited from participants in an institutionally funded cohort study, St. Jude Life, as well as from active ACT patients that meet eligibility criteria. The young adults in St. Jude Life are a highly motivated group who were followed in the After Completion of Therapy Clinic until age 18 years and a minimum of 10 years after their treatment ended if they were older than age 11 at the end of therapy
- Comparison Group: Potentially eligible comparison group participants will be recruited from the parent, older sibling, relative or friend population who accompany the ACT patient for follow-up at SJCRH. Parents (or siblings, relatives or friends who are 18 years or older) of children in remission, both from the active follow-up cohort (within five years of last treatment) and the After Completion of Therapy (ACT) cohort will be invited to complete the same assessments that the ALL survivor participants will complete. Comparison group participants are frequency matched to potentially eligible participants by race/ethnicity (white, black, other) age group (18 to 29, 30-39, 40-49 years) and gender.

SUMMARY:
The primary goal of this study is to provide comprehensive and objective information on impairments of musculoskeletal health, sensory function, and fitness among a large group of childhood ALL survivors, and to define high risk groups by assessing treatment factors that contribute to impaired function. This study includes a direct, objective evaluation of musculoskeletal function, sensory capacity, fitness, and physical activity patterns among adults who were treated for childhood ALL at St. Jude Children's Research Hospital (SJCRH) between 1980 and 1999. Among 899 ALL survivors, all of whom are eligible for an institutionally funded clinical study of medical late effects, the study will recruit 364 to participate in our evaluations. The study will also recruit 364 individuals for a comparison group, frequency matching on race/ethnicity, age and gender.

DETAILED DESCRIPTION:
The study will focus on the following primary objectives:

1. Enumerate the prevalence of musculoskeletal, sensory, and fitness impairments among adult survivors of childhood ALL. The study hypothesizes that adult survivors of childhood ALL will have a higher prevalence of musculoskeletal, sensory and fitness impairments than a control group frequency matched on race/ethnicity, age, and gender.
2. Evaluate the association between personal and treatment factors and musculoskeletal, sensory and fitness impairments. The study hypothesizes that:

   * Female gender, younger age at diagnosis, and cranial radiation will be associated with decreased lean body mass.
   * Female gender, younger age at diagnosis, and type of glucocorticoid (dexamethasone vs. prednisone) treatment will be associated with muscle weakness.
   * Sensory loss will vary as a function of age, with participants diagnosed at 12+ years of age demonstrating vincristine related sensory loss, and those diagnosed at <12 years of age demonstrating dexamethasone and/or intrathecal methotrexate related sensory loss.
   * Fitness impairments will be evident in participants who received 100 mg/m2+ of anthracyclines.

The study will focus on the secondary objectives:

1. Compare physical activity patterns between adult survivors of childhood ALL and a frequency matched control group. The study hypothesizes that adult survivors of childhood ALL will demonstrate lower levels of physical activity as measured with an activity monitor (accelerometer), and will report lower levels of overall physical activity, when compared to members of the comparison group.
2. Describe the association between habitual physical activity and energy expenditure among ALL survivors. The study hypothesizes that activity levels, measured with the accelerometer, will be positively correlated with energy expenditure, measured using the doubly labeled water technique.
3. Explore the associations between musculoskeletal and sensory health, and physical activity patterns among adult survivors of childhood ALL. The study hypothesizes that adult survivors of childhood ALL with lower proportions of lean muscle mass and/or sensory loss indicating peripheral neuropathy will demonstrate the lowest levels of physical activity.

ELIGIBILITY:
Inclusion Criteria:(ALL survivors):

1. Research participant who is a survivor of childhood ALL who was treated at St. Jude Children's Research Hospital between 1980 and 1999
2. Research participant must be at least ten years from diagnosis
3. Research participant must be at least 18 years of age at the time of the scheduled evaluation

Exclusion Criteria (ALL survivors):

1. Research participant who has Down Syndrome or congenital cognitive, musculoskeletal or cardiopulmonary impairments that interfere with motor function
2. Research participant currently pregnant or lactating
3. Research participant age 17 years or less
4. Research participant undergoing active treatment for cancer

Inclusion Criteria (Comparison Group)

1. Research participant is a sibling, parent, relative or friend of a current or former St. Jude patient.
2. Research participant must be at least 18 years of age at the time of the scheduled evaluation

Exclusion Criteria (Comparison Group)

1. Research participant who has Down Syndrome or congenital cognitive, musculoskeletal or cardiopulmonary impairments that interfere with motor function
2. Research participant currently pregnant or lactating
3. Research participant age 17 years or less
4. Research participant has a medical history of cancer
5. Research participant is a first degree relative of a survivor participating in MTRPAL

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study sample for this research will be recruited from participants in an institutionally funded cohort study, St. Jude Life, as well as from active ACT patients that meet eligibility criteria. The young adults in St. Jude Life are a highly motivated group who were followed in the After Completion of Therapy Clinic until age 18 years and a minimum of 10 years after their treatment ended if they were older than age 11 at the end of therapy. Potentially eligible comparison group participants will be recruited from the parent, older sibling, relative or friend population who accompany the ACT patient for follow-up at SJCRH. Parents (or siblings, relatives or friends who are 18 years or older) of children in remission, both from the active follow-up cohort (within five years of last treatment) and the After Completion of Therapy (ACT) cohort will be invited to complete the same assessments that the ALL survivor participants will complete.
Sampling Method: Probability Sample
Enrollment: 807 (Actual)
Dates: Start 2009-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Ascertain the prevalence of musculoskeletal, sensory, and fitness impairments among adult survivors of childhood ALL. | Day 1-2

SECONDARY OUTCOMES:
Compare physical activity patterns between adult survivors of childhood ALL and a frequency matched control group. | Day 1-7
Describe the association between habitual physical activity and energy expenditure among ALL survivors. | Day 1-7
Explore the associations between musculoskeletal and sensory health, and physical activity patterns among adult survivors of childhood ALL. | Day 1-7

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten K Ness, PT, Ph.D, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org